CLINICAL TRIAL: NCT04293783
Title: Efficacy of Lactobacillus Reuteri in Managing Social Deficits in Children With Autistic Spectrum Disorder: a Randomized Clinical Trial With Evaluation of Gut Microbiota and Metabolomics Profiles
Brief Title: Randomized Double-blind Clinical Trial With L.Reuteri Supplementation in Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Collaborators: University of Bari (Other)
Responsible Party: Principal Investigator, Luigi Mazzone, MD, PhD, University of Rome Tor Vergata
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Reg. Sperim. 244/19
Record Dates: First submitted 2020-02-26; First posted 2020-03-03 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Autism Spectrum Disorder
Keywords: Probiotic; Gut-Brain axis; L. Reuteri; Social Behavior; Microbiome; Metabolome; Inflammatory Profile; Gastrointestinal Symptoms
MeSH Terms: conditions — Autism Spectrum Disorder; Social Behavior

STUDY DESIGN:
Intervention Model Description: double-blind randomized, parallel-group, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Placebo chewable caps are identical in shape and taste to the test product, without the Lactobacillus reuteri components Both study products are delivered in identical containers and labelled as XXX.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L.Reuteri (Active Comparator): Lactobacillus reuteri DSM 17938 + Lactobacillus reuteri ATCC PTA 6475 two tablet by mouth 1 time per day
  Interventions: Dietary Supplement: L.Reuteri
- Placebo (Placebo Comparator): Placebo two tablet by mouth 1 times per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L.Reuteri — daily supplementation with two tablet for six months
  Other Names: Gastrus
  Arms: L.Reuteri
Dietary Supplement: Placebo — daily supplementation with two tablet for six months
  Arms: Placebo

SUMMARY:
The aim of this study is to assess the effects of a 6-months probiotic supplementation on behavioral profiles, microbiota and metabolic profiles, inflammatory biomarkers, gastrointestinal disturbances, in children with Autism Spectrum Disorders (ASD) with or without GI symptoms.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is a condition that includes social deficits, repetitive behaviors and language difficulties; its prevalence continues to increase worldwide, however, there are no medication for the core symptoms of this disorder. In addition to these core symptoms, children with ASD are 3.5 times more likely to suffer from gastrointestinal issues than children without developmental disorders. Moreover, GI problems have been associated with changes in the microbial communities inhabiting the gut of ASD individuals.

Studies in animal models have suggested that the gut microbes can modulate central nervous system-driven behaviors.

In 2019, a research group (Buffington et al.) found that a specific strain (L. Reuteri PTA) rescues the deficit in social interaction-induced VTA plasticity in ASD mouse, enhancing the salience and rewarding value of social stimuli.

These data support the idea that microbial therapies could ameliorate specific endophenotypes associates with ASD.

Aim of the study The aim of this pilot study is to determine the possible effects of supplementation with a specific probiotic strain (L. Reuteri ATCC PTA 6475) in ASD children on the core deficits of the disorder, the social behavior. A secondary aim is to evaluate the effects of probiotic supplementation on specific GI symptoms, and repetitive, dysfunctional behaviors, widely described in ASD children. Finally, the investigators will evaluate gut microbiota (fecal and salivary samples) and metabolomics (urinary samples) profiles differences before and after the supplementation.

Methods and participants Double blind randomized, placebo-controlled trial, with a nutritional supplement, with two parallel arms, an allocation ratio of 1:1, and a superiority framework.

The investigators aim to enroll 80 patients. A detailed informed consent will be given and and both parents will sign it before the start of the data collection.

The participants, after a first evaluation, will be divided into 2 groups; each arm will be blind randomized 1:1 to regular diet with a specific probiotic strain (L. Reuteri ATCC PTA 6475) or with placebo for 6 months.

After randomization the investigators will explain how to take the product and the first dose will be administered.

During the study the child is not allowed to take other probiotics. The type of neurologic/rehabilitation therapy ongoing at T0 cannot be changed until the study is finished.

Study Product Test product chewable tablets: 1x108 CFU Lactobacillus reuteri DSM 17938 + 1x108 CFU Lactobacillus reuteri ATCC PTA 6475 (together 2x108 CFU) Placebo chewable caps: identical in shape and taste to the test product without the Lactobacillus reuteri components Both study products are delivered in identical containers and labelled as XXX. Dosing: Two tablets/cps once a day.

Assessment

At the time of enrollment, each participant will undergo a comprehensive neuropsychological and biochemical evaluation, in order to establish the baseline of the primary and secondary outcome measures. A detailed Case Record Forms (CRF) containing all data pertinent to the study will be prepared.

At T0 the investigators will also collect blood, urinary salivary and fecal sample from each participant in order to perform biochemical, microbiological and metabolomics evaluation. The parents have to fill out questionnaire about dietary habits in a 5 day-diary.

After three months from the enrollment (T1), each child will undergo a second evaluation with some clinical and biological measures.

At the end of the study, six months from baseline, the investigators will perform another complete assessment through the same clinical, biochemical and neuropsychological evaluation performed at T0, to evaluate the possible changes in (1) autism symptoms severity; (2) affective and behavioral comorbid symptoms; (3) GI symptoms; (4) plasmatic, urinary and fecal biomarkers related to abnormal intestinal/inflammatory function. At T2, urinary salivary, and fecal sample will be also collected from each participant in order to perform microbiological and metabolomics evaluation.

All children recruited will undergo the evaluation at Child Neurology and Psychiatry unit, Policlinico Tor Vergata, Rome, Italy.

ELIGIBILITY:
Inclusion Criteria:

- Autism Spectrum Disorder (DSM-5 criteria diagnosis)

Exclusion Criteria:

* neurological syndromes (that explain autism symptoms)
* coeliac disease
* other organic GI disorder
* special diet.

Ages: 18 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Changes in severity level of ASD symptomatology | 6 months
  Delta of scores at Autism Diagnostic Observation Schedule-2
Changes in Microbiome Profile | 3 months and 6 months
  Characterization of the fecal and salivary microbiota by using a metagenomic approach (amplification and sequencing of a portion of the bacterial 16S rRNA) gene. A special focus is to evaluate if there is dysbiosis, if the supplementation rescues the dysbiosis and if these changes are correlated with the gastrointestinal and behavioral symptoms

SECONDARY OUTCOMES:
Changes in GI symptoms | 3 months and 6 months
  Delta of scores at GSRS (Gastrointestinal Symptoms Rating Scale). Higher scores are related to greater severity of symptoms
Changes in ASD symptomatology: problematic behaviors | 3 months and 6 months
  Delta of scores at ABC (Aberrant Behavior Checklist), a 58 item scale. Higher scores are related to greater severity of symptoms
Changes in ASD symptomatology: repetitive behaviors | 3 months and 6 months
  Delta of scores at RBS-R (Repetitive Behavior Scale-Revised), a 43 item scale. Higher scores are related to greater severity of symptoms
Changes in Adaptive Functioning | 6 months
  Delta of scores at Adaptive Behavior Assessment System-II
Changes in global ASD symptomatology | 3 months and 6 months
  Delta of scores at SRS (Social Responsiveness Scale). Higher scores are related to greater severity of symptoms
Changes in Behavioral Profiles | 3 months and 6 months
  Delta of scores at CBCL (Child Behavior CheckList)
Changes in Parental Stress | 3 months and 6 months
  Delta of scores at PSI (Parenting Stress Index)
Changes in Metabolomic Profile | 6 months
  Urinary samples collected for NMR analysis. Metabolomics profiles will be directed at biochemical processes such as neurotransmitter metabolism, gastrointestinal alterations or dysbiosis, and mitochondrial dysfunction). Furthermore, the effect of probiotic administration on the metabolome will be investigated.
Changes in Inflammatory Profile | 6 months
  Blood sample collected to evaluate changes in inflammatory profile (zonulin, IL-17 profile)

CONTACTS AND LOCATIONS:
Overall Officials: Mazzone Luigi, MD, PhD, Principal Investigator — University of Rome Tor Vergata; Francavilla Ruggiero, MD, PhD, Principal Investigator — University of Bari
Locations (2):
- Italy (2):
  - University of Bari, Bari, BA
  - University of Rome Tor Vergata, Rome, RM

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting 6 months after publication

REFERENCES:
- [Background] Sgritta M, Dooling SW, Buffington SA, Momin EN, Francis MB, Britton RA, Costa-Mattioli M. Mechanisms Underlying Microbial-Mediated Changes in Social Behavior in Mouse Models of Autism Spectrum Disorder. Neuron. 2019 Jan 16;101(2):246-259.e6. doi: 10.1016/j.neuron.2018.11.018. Epub 2018 Dec 3. PMID 30522820
- [Background] Vuong HE, Yano JM, Fung TC, Hsiao EY. The Microbiome and Host Behavior. Annu Rev Neurosci. 2017 Jul 25;40:21-49. doi: 10.1146/annurev-neuro-072116-031347. Epub 2017 Mar 8. PMID 28301775
- [Background] Schieve LA, Gonzalez V, Boulet SL, Visser SN, Rice CE, Van Naarden Braun K, Boyle CA. Concurrent medical conditions and health care use and needs among children with learning and behavioral developmental disabilities, National Health Interview Survey, 2006-2010. Res Dev Disabil. 2012 Mar-Apr;33(2):467-76. doi: 10.1016/j.ridd.2011.10.008. Epub 2011 Nov 24. PMID 22119694
- [Background] Lussu M, Noto A, Masili A, Rinaldi AC, Dessi A, De Angelis M, De Giacomo A, Fanos V, Atzori L, Francavilla R. The urinary 1 H-NMR metabolomics profile of an italian autistic children population and their unaffected siblings. Autism Res. 2017 Jun;10(6):1058-1066. doi: 10.1002/aur.1748. Epub 2017 Mar 11. PMID 28296209
- [Background] Indrio F, Di Mauro A, Riezzo G, Civardi E, Intini C, Corvaglia L, Ballardini E, Bisceglia M, Cinquetti M, Brazzoduro E, Del Vecchio A, Tafuri S, Francavilla R. Prophylactic use of a probiotic in the prevention of colic, regurgitation, and functional constipation: a randomized clinical trial. JAMA Pediatr. 2014 Mar;168(3):228-33. doi: 10.1001/jamapediatrics.2013.4367. PMID 24424513
- [Derived] Mazzone L, Dooling SW, Volpe E, Uljarevic M, Waters JL, Sabatini A, Arturi L, Abate R, Riccioni A, Siracusano M, Pereira M, Engstrand L, Cristofori F, Adduce D, Francavilla R, Costa-Mattioli M, Hardan AY. Precision microbial intervention improves social behavior but not autism severity: A pilot double-blind randomized placebo-controlled trial. Cell Host Microbe. 2024 Jan 10;32(1):106-116.e6. doi: 10.1016/j.chom.2023.11.021. Epub 2023 Dec 18. PMID 38113884